CLINICAL TRIAL: NCT00826137
Title: Prebiotics in the Prevention of Antibiotic-associated Diarrhea in Children
Brief Title: Preventing Childhood Antibiotic-associated Diarrhea by Prebiotics
Acronym: WGAAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sor472908ctil
Record Dates: First submitted 2008-12-29; First posted 2009-01-21 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Antibiotic-Associated Diarrhea
Keywords: prebiotics; Antibiotic-associated diarrhea
MeSH Terms: interventions — Inulin; fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Treated with prebiotics.
  Interventions: Dietary Supplement: Inulin and fructo-oligosaccharides.
- B (Placebo Comparator): Placebo treated.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Inulin and fructo-oligosaccharides. — Supplement during antibiotic treatment+14 days.
  Other Names: Placebo is base powder of product with no oligosaccharides.
  Arms: A
Dietary Supplement: Placebo — Placebo is base powder of product with no oligosaccharides.
  Arms: B

SUMMARY:
Prospective randomized double-blind study on the effect of prebiotics (inulin and fructo-oligosaccharides) in the prevention of antibiotic-associated diarrhea in children.

DETAILED DESCRIPTION:
Group will get either the product or placebo blindly throughout antibiotic treatment with additional 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with acute infection.

Exclusion Criteria:

* Hypersensitivity to antibiotics, chronic illness.

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Prevention of diarrhea. | During antibiotic treatment+14 days

SECONDARY OUTCOMES:
Duration of diarrhea. | During antibiotic treatment+14 days

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Weizman, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel